CLINICAL TRIAL: NCT00005201
Title: Idiopathic Dilated Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1080; R01HL036879 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-05

CONDITIONS: Heart Diseases; Cardiomyopathy, Congestive
MeSH Terms: conditions — Heart Diseases; Cardiomyopathy, Dilated

SUMMARY:
To determine the familial occurrence and pathogenesis of idiopathic dilated cardiomyopathy.

DETAILED DESCRIPTION:
BACKGROUND:

In 1987 idiopathic dilated cardiomyopathy was a disorder of unknown cause that directly affected one or both cardiac ventricles in a diffuse or multifactorial fashion, and that produced heart failure, at least in some patients. Although a viral etiology had been proposed, dilated cardiomyopathy could be associated with numerous genetic and non-genetic diseases. However in 1987, the role of genetic factors was not known in humans. Although the condition was usually dismissed as sporadic, numerous families with multiple affected members have been observed.

The role of atrial natriuretic peptide levels in the pathogenesis or progression of idiopathic dilated cardiomyopathy was just beginning to be explored in 1987. Although Syrian hamster studies did not suggest a genetic deficiency as the primary cause of dilated cardiomyopathy in that model, it was thought possible that ANP production or levels were somehow involved in how the myocardium responds in idiopathic dilated cardiomyopathy patients.

DESIGN NARRATIVE:

Eligible patients were interviewed and asked whether any first-degree relatives were willing to participate. If family members participated, a three generation pedigree was constructed and first-degree relatives contacted. The relatives were interviewed for a medical history and medical records from other institutions were reviewed. Each family member had a brief cardiovascular examination, a 12-lead electrocardiogram and 2-dimensional, M-mode, and Doppler echocardiogram. Blood was drawn for determination of atrial natriuretic peptide (ANP) levels. The contributions of variability in age, sex, drug use, smoking, and other concomitants to variability in ANP and echocardiographic data were estimated. After removing these sources of variability, the strength of similarity among family members was assessed. The relative contributions of genes and shared environments to the similarity among family members were estimated.

Heterogeneity in the mean levels of echocardiographic indices and ANP levels, familial aggregation and etiology of aggregation were assessed between families with familial idiopathic dilated cardiomyopathy and families with non-familial idiopathic dilated cardiomyopathy.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1987-07; Study Completion 1992-06 (Actual)

REFERENCES:
- [Background] Michels VV, Moll PP, Miller FA, Tajik AJ, Chu JS, Driscoll DJ, Burnett JC, Rodeheffer RJ, Chesebro JH, Tazelaar HD. The frequency of familial dilated cardiomyopathy in a series of patients with idiopathic dilated cardiomyopathy. N Engl J Med. 1992 Jan 9;326(2):77-82. doi: 10.1056/NEJM199201093260201. PMID 1727235
- [Background] Michels VV, Moll PP, Rodeheffer RJ, Miller FA Jr, Tajik AJ, Burnett JC Jr, Driscoll DJ, Thibodeau SN, Ansari AA, Herskowitz A. Circulating heart autoantibodies in familial as compared with nonfamilial idiopathic dilated cardiomyopathy. Mayo Clin Proc. 1994 Jan;69(1):24-7. doi: 10.1016/s0025-6196(12)61607-3. PMID 8271845